CLINICAL TRIAL: NCT01178970
Title: The Effects of Lower Body Resistance Training on Balance and Fall Prevention in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Thomas Allen, DO, University of Oklahoma
Allocation: Randomized | Model: Single Group
Other Study IDs: OU IRB 14759
Record Dates: First submitted 2010-07-21; First posted 2010-08-10 (Estimated); Last update posted 2010-08-10 (Estimated); Status verified 2010-08

CONDITIONS: Fall Prevention
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Resistance training

SUMMARY:
The aim of the study is to prevent falls related to poor lower body strength adn balance in the elderly.

DETAILED DESCRIPTION:
The purpose of the study is to determine the effects of a structured lower body resistance training program on balance in an elderly population. Our hypothesis is that elderly adults will improve their balance following a structured lower body strength training program compared to those who do not engage in a lower body strength training program.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female adults 65 or older with physician consent to participate

Exclusion Criteria:

* Unable to obtain physician consent to participate

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-08; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Balance improvement | 8 weeks
  Measured by:
  Postural orthostatic hypotension test-blood pressure taken while sitting and standing.
  Balanced test with Biodex Balance System SD-a person's ability to maintain balance on an unstable surface.

CONTACTS AND LOCATIONS:
Locations (1):
- OU-Tulsa Family Medicine Clinic, Tulsa, Oklahoma, United States